CLINICAL TRIAL: NCT06028932
Title: A Phase II Evaluation of Sacituzumab Govitecan (IMMU-132), an Anti-Trop-2-SN-38 Antibody-drug Conjugate in Recurrent or Persistent Platinum-resistant Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancers
Brief Title: A Study of Sacituzumab Govitecan (IMMU-132) in Platinum-resistant Ovarian Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000036114; 000 (Other: yctg)
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab govitecan, 10 mg/kg (Experimental): Sacituzumab govitecan, 10 mg/kg for the first 2 weeks of 21-day cycle until progression or adverse effects prohibit further treatment
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — Sacituzumab govitecan will be administered at 10 mg/kg weekly as an infusion for 2 consecutive weeks (2 weekly doses plus 1 week without treatment represents a single 3 week cycle). Treatment can be continued without a rest period in the absence of progression of disease or unacceptable toxicity.
  Other Names: IMMU-132

SUMMARY:
This is a non-randomized Phase 2 study of sacituzumab govitecan (IMMU-132) in subjects with recurrent or persistent platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal cancers.

DETAILED DESCRIPTION:
This is an open-label, Phase 2 study designed to assess the clinical activity of sacituzumab govitecan in subjects with recurrent or persistent platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have platinum-resistant (i.e., platinum-free interval <6 months) recurrent or persistent histologically confirmed epithelial (non-mucinous) ovarian, fallopian tube, or primary peritoneal cancer. Patients may have serous, endometrioid, clear cell, (pure or mixed), or undifferentiated histology.

  * Must have availability of archival tumor tissue FFPE block for TROP-2 testing
* All patients must have measurable disease. Measurable disease is defined as lesions which can be measured by physical examination or by means of medical imaging techniques. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpation or plain x-ray, or ≥ 10 mm when measured by spiral CT and/or MRI. Ascites and pleural effusions are not to be considered measurable disease.
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST v1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented, or a biopsy is obtained to confirm persistence following completion of radiation therapy.
* After undergoing surgery, patients may be optimally or sub optimally debulked.
* Patients with measurable recurrent disease of any previous substage (I-IV) are eligible to enrollment.
* Patients must have adequate bone marrow function: WBC greater than or equal to 3,000/ul, Platelets greater than or equal to 75,000/ul, Neutrophils greater than or equal to 1500/ul.
* Patients must have adequate renal function: creatinine less than or equal to 2.0 mg/dL.
* Patients must have adequate hepatic function: bilirubin ≤ 1.5 institutional upper limit of normal, aspartate aminotransferase [AST], and alanine aminotransferase [ALT] ≤ 2.5 × IULN or ≤ 5 × IULN if known liver metastases
* Patients must have an ECOG performance status of 0 or 1.
* Patients must have signed an approved informed consent.
* Patients must be at least 2 weeks beyond prior treatment (chemotherapy, investigational drugs including small molecular inhibitors, endocrine therapy, immunotherapy and/or radiation therapy) or major surgery.
* Patients must be at least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids <20 mg prednisone or equivalent daily are permitted)
* Patients must have recovered from all acute toxicities to Grade 1 or less from adverse events due to a previously administered agent

  * Note: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study
  * Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients with recurrent disease may have received no more than 2 prior chemotherapies for treatment of the recurrent ovarian cancer.

  * Adjuvant ± neoadjuvant are considered one line of therapy
  * Maintenance therapy (eg, bevacizumab, PARP inhibitors) are considered as part of the preceding line of therapy (ie, not counted independently).
  * Therapy changed due to toxicity or allergy in the absence of progression will be considered as part of the same line (ie, not counted independently).
* Patients may have received prior immunotherapy therapy alone or in combination with chemotherapy. A 4-week washout period is required between prior immunotherapy treatment and first dose of sacituzumab govitecan.
* Patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the study entry and must agree to use protocol-specific method(s) of contraception. .
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Patients with a positive serum pregnancy test or women who are breastfeeding.
* Patients with known hypersensitivity to the study drug, its metabolites, or formulation excipient.
* Patients who require ongoing therapy with or prior use of any prohibited medication(s) such as UGT1A1 inhibitors.
* Have other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancers or carcinoma in situ of the cervix, are excluded if there is any evidence of other malignancy being present within the last 5 years.
* Patients with a significant history of cardiac disease within 6 months, i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure (NYHA classification III-IV) or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring antiarrhythmia therapy.
* Patients with known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months
* Patients with any unstable medical issue (including cardiac issues as above, active treatment for symptomatic pulmonary embolism, CVA, renal or hepatic insufficiency, and active infection/sepsis requiring IV antibiotics).
* Have known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking ≤20 mg/day of prednisone or its equivalent. All patients with carcinomatous meningitis are excluded regardless of clinical stability
* Patients who have an uncontrolled seizure disorder, or active neurological disease.
* Have known history of HIV-1 or 2 (or positive HIV-1/2 antibody) with detectable viral load OR taking medications that may interfere with SN-38 metabolism
* Have active HBV or HCV. In subjects with a history of HBV or HCV, subjects with a detectable viral load will be excluded.
* Known hemorrhagic diathesis or active bleeding disorder.
* Patients with Gilbert's disease
* Presence of bulky disease (defined as any single mass >7 cm in its greatest dimension). Patients with a mass over 7 cm, but otherwise eligible, may be considered for enrollment after discussion and approval with the study PI.
* Patients with active ≥ grade 2 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
* Prior history of clinically significant bleeding, intestinal obstruction, or GI perforation within 6 months of initiation of study treatment.
* Patients with a history of an anaphylactic reaction to irinotecan or ≥ Grade 3 GI toxicity to prior irinotecan.
* Have previously received topoisomerase I inhibitors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 4 Years
  Objective response rate (complete response and partial response rates) by RECIST1.1 criteria in patients with platinum resistant recurrent ovarian carcinoma.

SECONDARY OUTCOMES:
Duration of overall survival (OS) | 6 Years
  Overall survival is defined as the duration of time from study entry to death or the date of last contact.
Duration of progression free survival (PFS) | 6 Years
  Progression free survival is defined as the duration of time from study entry to time of progression, death, or is censored at date of last disease assessment
Durable disease control rate (DDCR) | 6 Years
  The percentage of patients who have achieved complete response, partial response, and stable disease.
Assess the safety profile of sacituzumab govitecan in ovarian cancer patients (adverse events as assessed by CTCAE v5.0) | 6 Years
  Incidence of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Santin, M.D., Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greenman M, Bellone S, Demirkiran C, Max Philipp Hartwich T, Santin AD. Sacituzumab govitecan in heavily pretreated, platinum-resistant high grade serous ovarian cancer. Gynecol Oncol Rep. 2024 Jul 13;54:101459. doi: 10.1016/j.gore.2024.101459. eCollection 2024 Aug. PMID 39108617